CLINICAL TRIAL: NCT07217444
Title: Improving Outcomes in Adolescent Inpatient Depression With Deep Transcranial Magnetic Stimulation
Acronym: IMPACT-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Rana Elmaghraby, ASSISTANT PROFESSOR, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-0385
Record Dates: First submitted 2025-10-08; First posted 2025-10-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder (MDD); Suicidal Ideation; Hospitalization in Children
Keywords: Major Depressive Disorder; MDD; Transcranial Magnetic Stimulation (TMS); Deep Transcranial Magnetic Stimulation; dTMS
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: It's a randomized sham-controlled trial with deep Transcranial Magnetic Stimulation (dTMS) treatment and sham controlled group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active dTMS Treatment (Active Comparator): Participants will receive active dTMS 5 sessions per day for 5 days
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham controlled (Sham Comparator): Sham dTMS 5 sessions per day for 5 days. If participants in the sham group do not show a significant treatment response by the 12th month follow-up -reduction in depression symptoms from screening - they will then become eligible for and offered active, open-label treatment.
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The Brainsway Deep TMS System with the FDA-cleared H7 Coil will be used to deliver all accelerated theta burst stimulation (aTBS) sessions. The H7 Coil is designed to target deeper and broader brain regions, including the prefrontal and anterior cingulate cortices, and has FDA 510(k) clearance for treatment of OCD and MDD in adults. Stimulation will follow a standardized accelerated theta burst protocol: triplet 50 Hz bursts delivered every 200 ms (5 Hz), in 2-second trains with 8 seconds off, at 90% RMT, totaling 600 pulses per session. Participants will receive five sessions per day over five business days with 30-minute breaks between the third and fourth sessions and exceeding or preceding these breaks will not be a protocol deviation. The sham coil mimics sensory experience without delivering stimulation.
  Arms: Active dTMS Treatment
Device: Transcranial Magnetic Stimulation Sham — Investigators will use a robust sham technique that is manufacturer-designed to mimic the auditory and tactile sensations of active TMS without delivering effective magnetic stimulation to the brain. The Brainsway Sham H7-CoilTM will be utilized for treatment delivery. The H-7 coil already has a built-in sham system that can operate as a placebo. Only the TMS operators will have access to intervention assignments, the rest of the study team will not have access to assignments to maintain the blinded status of participants, caregivers, and raters.
  Arms: Sham controlled

SUMMARY:
Evaluate the feasibility, safety, and preliminary efficacy of deep Transcranial Magnetic Stimulation (dTMS) as an adjunctive treatment for adolescents hospitalized with major depressive disorder (MDD).

DETAILED DESCRIPTION:
The overall goal of this study is to evaluate the feasibility, safety, and preliminary efficacy of deep Transcranial Magnetic Stimulation (dTMS) as an adjunctive treatment for adolescents hospitalized with major depressive disorder (MDD). Our central hypotheses are that dTMS H7 targeting the dorsomedial prefrontal and cingulate cortices, delivered via the Brainsway H7-Coil™, will be safe, well tolerated, and lead to improved depressive symptoms, reduced suicide risk, and lower readmission rates compared to sham treatment. Investigators propose a double-blind, sham-controlled randomized clinical trial enrolling 14- to 18-year-old inpatients with MDD with or without obsessive compulsive disorder (OCD). Participants (n=60) will be randomized to receive either active or sham TMS during hospitalization, with follow-up assessments continuing for 12 months post-discharge. Outcomes will include safety, tolerability, treatment adherence, depressive symptom change, suicidal ideation, and time to psychiatric readmission. This study will provide foundational data to support the clinical integration of TMS into inpatient care for adolescents with treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English and able to volunteer in the informed consent process and provide spontaneous narrative description of key elements, risks, and benefits of the study.
2. Aged 14 years to 18 years, inclusive.
3. Diagnosis of MDD based on psychologist diagnosis and DSM-5-checklist based interview.
4. Symptoms of moderate to severe depression according to Hamilton Depression Rating Scale Score > 20.
5. Participants are not required to discontinue current interventions

Exclusion Criteria:

1. Participation in an investigational drug trial within the past three months.
2. Contraindications to Transcranial Magnetic Stimulation including, but not limited to, a history of epilepsy, the presence of metallic foreign bodies, or implanted medical devices (e.g. ventriculoperitoneal shunt, pacemaker, medical pump).
3. Actively psychotic (i.e. disorganized, delusional, paranoid, or having hallucinations)
4. Actively suicidal (have a suicidal plan and intent and is on 1:1 close observation)
5. For female subjects of childbearing potential, a positive urine pregnancy test.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Tolerability and Safety | Completed before and immediately after the intervention
  We will collect and summarize descriptive data on discomfort and adverse events using Sections IV of the TMS Adverse Events and Associated Sensations Questionnaire (TMSens_Q). This captures typical sensory experiences or side effects, e.g. scalp tingling or headache) as well as adverse events (e.g. syncope). Tolerability will be characterized based on sensory experiences and side effects, comparing active to sham treatment. Safety will be further assessed by the rate of early discontinuation due to intolerability or adverse events using the CCHMC Adverse Event form.
  Tolerability:
  Unit of measure: frequency and severity of sensory experiences and adverse events, e.g. scalp tingling or headache, syncope).
  Safety:
  Unit of measure: Rate of early discontinuation or withdrawal of treatment due to intolerability or adverse events.

SECONDARY OUTCOMES:
Hospitalization | Completed monthly for the first 6 months, 9th and 12th month follow up
  Time to first psychiatric readmission or emergency department (ED) visit for depression or suicidality within 12 months post-discharge.
  Unit of Measure: Time to first psychiatric readmission or ED visit (months).
Depression Symptoms | Completed at screening, same day after the intervention, monthly for 6 months, then at 9th and 12th month follow up
  Change in depressive symptom severity as rated by the Hamilton Depression Rating Scale (HDRS-17). The HDRS is a 17-item rating scale administered by a trained rater following a semi-structured interview. Scores of 0-7 are generally within the normal range, and a score of 20 or higher indicates moderate depression severity. Research suggests that a decrement of 7 points on the HAMD-17 represents minimally clinically important differences from patient perspectives.
  Unit of Measure:
  HDRS-17 total score.
Suicide Risk | Completed at screening, same day after the intervention, monthly for 6 months, then at 9th and 12th month follow up
  Change in suicidal ideation and behavior from screening to follow-up, assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS).
  Unit of Measure:
  C-SSRS severity.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Elmaghraby, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All the IPD collected throughout this trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the completion of data collection